CLINICAL TRIAL: NCT00881101
Title: Dose Escalation Study of Liposomal Paclitaxel in Chinese Patients With Advanced Solid Tumors
Brief Title: Clinical Study of Liposomal Paclitaxel in Chinese Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing Sike Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Jin Li, Dr., Cancer Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS- PH I -01-2009
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Solid Tumor
Keywords: Liposomal Paclitaxel; Maximum tolerated dose; Dose limiting toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Liposomal paclitaxel
  Interventions: Drug: Liposomal paclitaxel

INTERVENTIONS:
Drug: Liposomal paclitaxel — All Patients will receive liposomal paclitaxel (starting at a dose of 190mg/m2,3h,ivgtt,at d1)each cycle for 1 cycle.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and dose limiting toxicities of liposomal paclitaxel in Chinese patients with solid tumors in advanced stages.

DETAILED DESCRIPTION:
There are clinical trials show that paclitaxel is common option for the treatment of solid tumors. Liposomal paclitaxel has different pharmacokinetic features comparing with conventional paclitaxel. However,the tolerance of this new dosage form of paclitaxel (liposomal paclitaxel) has never been studied in Chinese cancer patients. This study is designed to find the maximum tolerated dose and dose limiting toxicities of liposomal paclitaxel in Chinese cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: from 18 to 70
2. Patients with solid tuomors at advanced stage must be histologically or cytologically confirmed ,and be suitable for treating with Paclitaxel Liposome solo
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS)is from 0 to 2
4. Patients who are expected to live at least 3 months
5. Laboratory tests before the study: white blood count (WBC)≥4,000/mm³,absolute neutrophil count (ANC) ≥1,500/mm³, platelet count ≥100,000/mm³, hemoglobin≥9.0 g/dL, aspartate aminotransferase AST (sGOT) and alanine aminotransferase ALT(sGPT)≤2.5 times of normal value upper limit，serum creatinine≤1.0 time of normal value upper limit，total bilirubin≤1.5 times of normal value upper limit
6. Not using chemotherapeutics (including test drug)before the study trial at least 4 weeks
7. No obvious functional disturbance diseases of internal organs
8. Complying with the study protocol
9. Sign informed consent
10. No Previous anaphylactic reaction to hormone

Exclusion Criteria:

1. Allergy to any medication or foods; History of hypersensitivity reactions to the conventional dosage form of paclitaxel or correlate excipients
2. Active uncontrolled central nervous system metastasis
3. Severe complications that obviously influence the compliance of patients
4. Grade ≥1 neuropathy using NCI CTCAE version 3.0 criteria
5. Taking other study medications or participating other clinical trial within 4w
6. Having radiation therapy or operation within 4w
7. Any non-remission toxicity ≥ CTC 1 in prior anticancer therapy(including radiation therapy) (except alopecie and hemoglobin)
8. Pregnant or lactant women; fertile patients not using effective contraception during study
9. No chief organ functional disturbance or diseases:

   * abnormal liver and renal functions
   * myocardial infarction
   * active heart disease
   * neuropathy or mental diseases including dementia or epilepsy
   * blind、deaf、dumb or extremity disability
   * known infection
   * active diffuse intravascular coagulation
10. Others whom researchers regard not eligible for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose | 6 months

SECONDARY OUTCOMES:
dose limiting toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Dr., Principal Investigator — Cancer Hospital of Fudan University
Locations (1):
- The ethics committee of Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality, China